CLINICAL TRIAL: NCT07010549
Title: Clinical and Instrumental Evaluation of the Face Biorevitalization Effect With the Medical Device Foliage Hydrofil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phitogen Beauty Labs SRL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLIAGE-2022
Record Dates: First submitted 2025-03-20; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Skin Ageing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm for evaluation of the skin hydration modification from baseline to Day 98. (Experimental): Each treatment session will involve multiple microinjections, with needles 30G 4mm, in the face (external corner of the eye and cheek). The amount of product injected will be up to 2 mL, according to Investigator's judgement; the microinjections will be performed at a distance of 1-2 cm from each other. An anesthetic cream could be used before injections, at Investigator's discretion.
  Interventions: Device: Hyaluronic Acid injections

INTERVENTIONS:
Device: Hyaluronic Acid injections — Among treatments today available, bio-revitalization is a process which triggers the skin's own, natural collagen production and cell rejuvenation through the injection of hyaluronic acid serums. This substance is hydrophilic, drawing many times its weight in water. As we age, we have less naturally produced HA in our tissues and skin dehydration becomes a telltale sign of aging. The HA owns a great hydrating power, due to this property is widely used in the biorevitalization treatments. Its use results in supple, younger-looking skin with reduced wrinkles and improved elasticity.In bio-revitalization procedures that involve intradermal micro-injections of natural HA, with a molecular weight close to the endogenous one, carried out in correspondence with the imperfections, the viscoelastic properties of HA allow to rehydrate the tissues, allowing to prevent and contrast the aging process skin and promote their remodeling.

SUMMARY:
this is a Post market, prospective, single arm, clinical investigation. Foliage Hydrofil is a CE marked, class III, resorbable medical device (sterile, non-pyrogenic and physiological gel) to be used for the hydration of the skin and for the correction of superficial skin imperfections of the face and body and in the process of repairing the dermal tissue. The main component of Foliage Hydrofil is HA sodium salt of non-animal origin, produced by bacterial fermentation. Each subject will receive three treatments, one vial 2mL (1.6% HA formulation) each, with Foliage Hydrofil, 3 weeks apart. Foliage Hydrofil will be injected with needles 30G 4mm only. The area treated with the study treatment will be the face. The device administration could be done after an anesthetic cream application, according to Investigator's judgement.

Primary objective

* To evaluate the clinical performance of Foliage Hydrofil in the improvement of the skin hydration in the treated area (face) at Day 98, from baseline. Secondary objectives
* To evaluate the clinical performance of Foliage Hydrofil in the improvement of the skin hydration in the treated area at Day 21 and 42, from baseline;
* To evaluate the improvement of the skin texture, skin tone, smoothing of fine lines and wrinkles in the treated area at Day 21, 42 and 98, from baseline;
* To evaluate the aesthetic change from baseline as judged by the Investigator at Day 21, 42 and 98;
* To evaluate the aesthetic change from baseline as judged by the subject at Day 21, 42 and 98;
* To evaluate the subject's satisfaction at Day 21, 42 and 98

Safety objectives

* To assess the local safety at injection site (pain, erythema, edema, bruising) of the treatment with Foliage Hydrofil;
* To assess the systemic safety of the treatment with Foliage Hydrofil.

DETAILED DESCRIPTION:
Study Visits and Assessments

Visit 1 screening - baseline- treatment start (day 1):

Subjects will be evaluated with regard to the inclusion and exclusion criteria that will allow their participation into the study. Before any study specific evaluation is carried out, subjects will receive all the information about the study by the Investigator and will sign an informed consent form.

The following activities will be performed at first visit:

* Collection of demographic information
* Medical and surgical history
* Physical examination (focused on the skin)
* Previous (in the 30 days before) and concomitant medications / treatments recording
* Urine pregnancy test (where applicable)
* Inclusion/exclusion criteria assessment
* Photos of the treated area (before injections)
* Corneometer examination of treated area (before injections)
* Skin surface characteristics, texture, tone, fine lines and wrinkles (before injections)
* First treatment
* Local and systemic adverse events after the first treatment. The following treatment session will be scheduled three weeks later, with a window of ± 4 days. The subject will be solicited to contact the Investigator for any problem between visits.

Visit 2 (Day 21 ± 4) and Visit 3 (Day 42 ± 4):

The following activities will be done at Visit 2, and 3:

* Physical examination (focused on the skin)
* Change in concomitant medications / treatments recording
* Photos of the treated area (before second/third injection session)
* Corneometer examination of treated area (before second/third injection session)
* Skin surface characteristics, texture, tone, fine lines and wrinkles (before second/third injection session)
* PAIS Subject
* GAIS Investigator
* Second/third treatment
* Adverse events (occurred since previous visit) recording
* Local and systemic adverse events after the second/third treatment. The second and third treatment sessions will be scheduled three weeks apart from each other, with a window of ± 4 days. The subject will be solicited to contact the Investigator for any problem between visits. The final visit will be scheduled about 2 months after last treatment session.

Visit 4 - End of study (Day 98 ±7):

The following activities will be done at Visit 4:

* Physical examination (focused on the skin)
* Change in concomitant medications / treatments recording
* Photos of the treated area
* Corneometer examination of treated area
* Skin surface characteristics, texture, tone, fine lines and wrinkles
* PAIS Subject
* GAIS Investigator
* Overall satisfaction by subject
* Adverse events (occurred since previous visit) recording. Should the subject interrupt or conclude in advance the clinical study, for any reason, a Visit 4 will be completed

ELIGIBILITY:
Inclusion Criteria:

Subjects presenting all the following inclusion criteria will be eligible to enter the study:

1. Generally healthy man and women, aged between 30 and 55 years (inclusive), looking for aesthetic procedures to improve the aspect of their face.
2. Caucasian race (skin type from I to IV as per Fitzpatrick Skin Type scale)
3. Visible signs of skin aging in the face (e.g. reduced skin elasticity, reduced turgor, actinic elastosis, smaller and larger wrinkles) according to the Investigators opinion;
4. Corneometer Capacitance of the area treated < 80
5. Subjects wishing not to modify their lifestyle during the study period;
6. Subjects with cooperative attitude, able to comprehend the full nature and the purpose of the investigation, including possible risks, side effects and discomforts and willing to adhere to the study schedule (including attendance to the planned visits) and study prescriptions;
7. Written informed consent release prior to any study-related procedures. -

Exclusion Criteria:

Subjects presenting one or more of the following exclusion criteria will not be eligible to enter the study:

1. Pregnancy or breastfeeding woman or woman of childbearing potential not practicing adequate contraception.
2. Subjects with Fitzpatrick skin type from V to VI
3. Subjects with known allergy/hypersensitivity to product components.
4. Extensively photo damaged and aged skin according to the Investigators opinion.
5. Active skin disease, inflammation or related conditions, such as infection, perioral dermatitis, seborrheic eczema and rosacea in the face, hands or décolletage.
6. Immune system disorders
7. History of or active collagenosis (e.g. systemic lupus, erythematosis, rheumatic arthritis, skin or systemic sclerosis).
8. Concomitant therapy with thrombolytics or anticoagulants, or have taken inhibitors of platelet aggregation, within 2 weeks before the first product administration.
9. History of cancerous or pre-cancerous lesions in the face, neck and décolletage.
10. Tattoo/s on the skin around the treatment site
11. Previous tissue augmenting therapy with non-permanent filler or treatment with botulinum toxin, aesthetic surgical therapy, laser treatment, mesotherapy, or any form of peeling in the face, hands or décolletage within 12 months prior to the baseline visit.
12. Use of injectable revitalization preparations within 12 months prior to the baseline visit.
13. Use of retinoic acid within 6 months prior to the baseline visit.
14. Previous or concomitant treatment with chemotherapy, immunosuppressive agents or corticoids.
15. History of treatment with permanent filling materials.
16. Participation in any other clinical study within 30 days prior to the first visit or plan to participate in another clinical study during this study period.
17. Planned or ongoing weight reduction program during the study.
18. Known history of drug or alcohol abuse within 6 months prior to the baseline visit.
19. Known hypersensitivity to one or more components of anesthetic creams
20. Nicotine use during the study or stopped within 12 months before the first visit.
21. Any medical condition that in the opinion of the Investigator makes the subject unsuitable for inclusion (e.g. severe chronic disease, malignancy, bleeding disorder, skin diseases etc).
22. Other condition preventing the subject to entering the study in the Investigator's opinion e.g. subjects anticipated to be unreliable, unable to return for the follow-up visits, not likely to avoid other prohibited treatments or procedures or incapable of understanding the information or instructions. -

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical performance of Foliage Hydrofil in the improvement of the skin hydration in the treated area (face) at Day 98, from baseline | day 98
  The primary endpoint of the study is the change in skin hydration from baseline to Day 98, evaluated through corneometer skin examination.

SECONDARY OUTCOMES:
clinical performance of Foliage Hydrofil in the change of the skin hydration in the treated area at Day 21 42, from baseline | day 21 - day 42
  the evaluation of the change in skin hydration from baseline to Day 21 and 42, through corneometer examination.
subject overall satisfaction | Day 21, 42 and 98
  The subject will be asked "Please express your degree of satisfaction with the treatment received" through a 5-points scale (1 very much satisfied, 2 satisfied,3 not satisfied nor unsatisfied, 4 unsatisfied, 5 very unsatisfied).
skin texture changement | Day 21, 42 and 98
  the investigator will evaluate in his or her own judgment the skin texture as follows: poor-good-very good
Investigator's assessment | Day 21, 42 and 98
  the Investigator's aesthetic change assessment using the Global Aesthetic Improvement Scale (GAIS) as follows:
  1. worse tha before treatment
  2. no change
  3. minimal improvement
  4. good improvement
  5. optimal improvement
subject's assessment | Day 21, 42 and 98
  the subject's aesthetic change assessment using the Patient's Aesthetic Improvement Scale (PAIS) as follows:
  1. worse
  2. no change
  3. somewhat improved
  4. moderately improved
  5. very much improved
Smoothing of fine lines | Day 21, 42 and 98
  the investigator will evaluate in his or her own judgment the smoothing of fine lines as follows: poor-good-very good
skin tone changement | Day 21, 42 and 98
  the investigator will evaluate in his or her own judgment the skin tone as follows: poor-sufficient-middle-good
Wrinkles modification | Day 21, 42 and 98
  the investigator will evaluate in his or her own judgment the wrinkles modification as follows:
  1. absent
  2. slight
  3. Moderate
  4. Severe
  5. Extreme

CONTACTS AND LOCATIONS:
Overall Officials: Tiziana Lazzari, Principal Investigator — Poliambulatorio di Medicina Estetica Casa della Salute SPA Largo XII Ottobre, 62 16121 GENOVA
Locations (1):
- Poliambulatorio di Medicina Estetica Casa della Salute SPA, Largo XII Ottobre, 62, Genova, Italy

REFERENCES:
- [Derived] Chahine S, Marozzi B, Valle A, Michellini L, Lazzari T. Efficacy and Safety of Non-cross-Linked Hyaluronic Acid Injections for Facial Skin Biorevitalization: A Single-Center, Open-Label, Single-Arm, Uncontrolled, Post-marketing Study. Cureus. 2025 Aug 13;17(8):e90005. doi: 10.7759/cureus.90005. eCollection 2025 Aug. PMID 40951208

DOCUMENTS (4):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT07010549/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT07010549/SAP_001.pdf
  • Informed Consent Form: informed consent (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT07010549/ICF_002.pdf
  • Informed Consent Form: information sheet (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT07010549/ICF_003.pdf